CLINICAL TRIAL: NCT02539186
Title: The Effect of Sono-guided Injection With Platelet Rich Plasma for Carpal Tunnel Syndrome
Brief Title: The Effect of Platelet Rich Plasma for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB No: 1-104-05-108
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet rich plasma (Experimental): Sono-guided injection with 3cc platelet rich plasma between carpal tunnel and median nerve in intervention group.
  Interventions: Biological: platelet rich plasma
- splinting (Active Comparator): The wrist night splint was firmly fixed in a neutral position to immobilize the affected wrist. Patients were ordered to wear the splint while resting at night and at least 8 hours per day during the period of study in control group.
  Interventions: Device: splint

INTERVENTIONS:
Biological: platelet rich plasma — Sono-guided injection with 3cc platelet rich plasma between carpal tunnel and median nerve
  Arms: platelet rich plasma
Device: splint
  Arms: splinting

SUMMARY:
The platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders. Although few studies have showed beneficial effect of PRP for regeneration of peripheral neuropathy in animal study, the associated study in human is rare.

DETAILED DESCRIPTION:
The platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders. Although few studies have showed beneficial effect of PRP for regeneration of peripheral neuropathy in animal study, the associated study in human is rare. We performe a prospective study to investigate the effect of PRP in patients with carpal tunnel syndrome.

Patients with carpal tunnel syndrome (CTS) were randomized into intervention and control group. Participants in intervention group received sono-guided injection with 3cc PRP and control group received night splint. The evaluation was performed pretreatment as well as on the 1st, 4th, 8th, 12th, 16th and 24 week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 year-old.
2. Typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test, numbness/tingling in at least two of the first, second, or third digits, and in whom the diagnosis was confirmed using an electrophysiological study.

Exclusion Criteria:

1. Cancer
2. Coagulopathy
3. Pregnancy
4. Inflammation status
5. Patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previously undergone wrist surgery or steroid injection for CTS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Change from baseline of severity of symptoms and functional status 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline of cross-sectional area in median nerve on 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline of electrophysiological study on 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  electrophysiological study according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA).
Change from baseline in finger pinch on 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 1st, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  The finger pinch strength was measured using Jamar dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, School of Medicine, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan

REFERENCES:
- [Background] Kucuk L, Gunay H, Erbas O, Kucuk U, Atamaz F, Coskunol E. Effects of platelet-rich plasma on nerve regeneration in a rat model. Acta Orthop Traumatol Turc. 2014;48(4):449-54. doi: 10.3944/AOTT.2014.13.0029. PMID 25230270
- [Background] Zheng C, Zhu Q, Liu X, Huang X, He C, Jiang L, Quan D, Zhou X, Zhu Z. Effect of platelet-rich plasma (PRP) concentration on proliferation, neurotrophic function and migration of Schwann cells in vitro. J Tissue Eng Regen Med. 2016 May;10(5):428-36. doi: 10.1002/term.1756. Epub 2013 May 31. PMID 23723151
- [Background] Lichtenfels M, Colome L, Sebben AD, Braga-Silva J. Effect of Platelet Rich Plasma and Platelet Rich Fibrin on sciatic nerve regeneration in a rat model. Microsurgery. 2013 Jul;33(5):383-90. doi: 10.1002/micr.22105. Epub 2013 May 2. PMID 23640879
- [Background] Park GY, Kwon DR. Platelet-rich plasma limits the nerve injury caused by 10% dextrose in the rabbit median nerve. Muscle Nerve. 2014 Jan;49(1):56-60. doi: 10.1002/mus.23863. Epub 2013 Sep 20. PMID 23558771